CLINICAL TRIAL: NCT03207958
Title: A Pilot Study of Belimumab (Benlysta) for Prevention of Chronic Graft-versus-Host Disease Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: Belimumab for Prevention of Chronic Graft-versus-Host Disease Following Allogeneic Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: GlaxoSmithKline (Industry); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201709068
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Graft Vs Host Disease; Graft-versus-host-disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Belimumab (Experimental): * Subjects meeting eligibility criteria will start treatment between Day +3- and Day +60 after alloHCT
  * Belimumab will be administered intravenously every 2 weeks for 3 cycles and then every 4 weeks for a total of 7 cycles (6 months)
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — -Given over 1 hour
  Other Names: Benlysta

SUMMARY:
Given the role of B cells in the pathophysiology of chronic graft versus host disease (GvHD), the association between elevated BAFF levels post-transplant in abnormal B-cell homeostasis and chronic GvHD, and the efficacy of belimumab in the inhibition of soluble human B lymphocyte stimulator protein (BAFF) signaling, these proof-of-principle findings support the rational for use of belimumab as prophylaxis of chronic GvHD. The investigators propose a pilot and feasibility study to assess the safety and tolerability, as well as preliminary efficacy, of belimumab as prophylaxis of chronic GvHD following allogeneic hematopoietic cell transplantation (alloHCT). The investigators' central hypothesis is that belimumab will be well tolerated and have a favorable effect on incidence and severity of chronic GvHD.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Diagnosis of hematologic malignancy (i.e. acute myeloid leukemia, acute lymphoblastic leukemia, chronic lymphocytic leukemia, chronic myelogenous leukemia, Hodgkin's lymphoma, non-Hodgkin's lymphoma, myelodysplastic syndrome, chronic myelomonocytic leukemia)
* Use of myeloablative or non-myeloablative conditioning regimen
* Use of mobilized peripheral blood stem cells from fully HLA-matched related or unrelated donor as a graft source
* Acute GvHD prophylaxis with methotrexate and tacrolimus
* Documented complete remission with full donor engraftment (by STR identity testing) on Day +30 bone marrow biopsy

  * Complete remission: less than 5% blasts in an aspirate bone marrow sample with a count of at least 200 nucleated cells, no blasts with Auer rods or persistence of extramedullary disease PLUS absolute neutrophil count (ANC) > 1,500/μL, platelet count ≥ 50,000/μL and no leukemic blasts in the peripheral blood.
  * Negative minimal residual disease
  * Full donor engraftment by STR testing (either by bone marrow or peripheral blood testing)
* Adequate end organ function:

  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
  * Creatinine clearance ≥ 40 mL/min/1.73 m^2 by the Cockcroft-Gault formula
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 16 weeks after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an Institutional Review Board (IRB)-approved written informed consent.

Exclusion Criteria:

* Active grade III-IV classic acute GvHD; subjects with prior resolved acute GvHD on stable doses of immunosuppression at time of enrollment will be permitted
* Evidence of classic chronic GvHD or overlap chronic GvHD at time of enrollment
* Subjects who participated in a clinical trial of acute GvHD prophylaxis in which chronic GvHD was a secondary end point
* Donor lymphocyte infusion administered to treat relapse or loss of donor chimerism
* Treatment with rituximab or other anti-B cell specific antibodies within previous 3 months
* History of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix
* Currently receiving any other investigational agents
* Known allergy or intolerance to any component of belimumab, including human or murine proteins or monoclonal antibodies
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations (including current drug or alcohol abuse or dependence, or history of drug or alcohol abuse or dependence within the last year) that would limit compliance with study requirements
* Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 14 days prior to planned start of therapy
* Evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months and/or poses a significant suicide risk in the judgment of the investigator
* History of pre-existing immunodeficiency disorder, autoimmune condition, or chronic infection
* Known HIV positivity
* Serologic evidence of current or past hepatitis B infection based on the results of testing for HBsAg and anti-HBc - Patients positive for HBsAg or HBcAb are excluded
* Positive test for hepatitis C antibody (patients with documented clearance of hepatitis C by PCR following treatment will be permitted)
* Currently on therapy for active chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria). Prophylactic therapy is allowed.
* Has any other clinically significant abnormal laboratory value in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of belimumab as prophylaxis of chronic GvHD in subjects following alloHCT as measured by number of participants who experience each adverse event | 30 days following the completion of treatment (approximately 7 months)
  -Adverse events will be graded according to CTCAE v4.03.

SECONDARY OUTCOMES:
Incidence and severity of chronic GvHD | 6 months after alloHCT
  -The presence of chronic GvHD will be determined according to the 2014 NIH Criteria. If chronic GvHD is diagnosed, each organ will be scored 0-3 and graded, according to the 2014 NIH criteria for Diagnosing and Staging of Chronic GvHD. These data will allow calculation of the NIH global severity score of mild, moderate or severe.
Incidence and severity of chronic GvHD | 12 months after alloHCT
  -The presence of chronic GvHD will be determined according to the 2014 NIH Criteria. If chronic GvHD is diagnosed, each organ will be scored 0-3 and graded, according to the 2014 NIH criteria for Diagnosing and Staging of Chronic GvHD. These data will allow calculation of the NIH global severity score of mild, moderate or severe.
Incidence and severity of chronic GvHD | 24 months after alloHCT
  -The presence of chronic GvHD will be determined according to the 2014 NIH Criteria. If chronic GvHD is diagnosed, each organ will be scored 0-3 and graded, according to the 2014 NIH criteria for Diagnosing and Staging of Chronic GvHD. These data will allow calculation of the NIH global severity score of mild, moderate or severe.
Incidence and severity of acute GvHD | 3 months after alloHCT
  -Acute GvHD will be graded according to modified Glucksberg scale (I-IV)
Incidence and severity of acute GvHD | 6 months after alloHCT
  -Acute GvHD will be graded according to modified Glucksberg scale (I-IV)
Overall survival | 6 months after alloHCT
  -Overall survival will be determined from date of belimumab initiation, with death from any cause as the event of interest, and censoring at last follow up date for those with incomplete observations.
Overall survival | 12 months after alloHCT
  -Overall survival will be determined from date of belimumab initiation, with death from any cause as the event of interest, and censoring at last follow up date for those with incomplete observations.
Overall survival | 24 months after alloHCT
  -Overall survival will be determined from date of belimumab initiation, with death from any cause as the event of interest, and censoring at last follow up date for those with incomplete observations.
Relapse rate | 6 months after alloHCT
  -Relapse rate will be determined from date of belimumab initiation and censoring at last follow up date for those with incomplete observations.
Relapse rate | 12 months after alloHCT
  -Relapse rate will be determined from date of belimumab initiation and censoring at last follow up date for those with incomplete observations.
Relapse rate | 24 months after alloHCT
  -Relapse rate will be determined from date of belimumab initiation and censoring at last follow up date for those with incomplete observations.
Overall corticosteroid requirement for treatment of chronic GvHD as measured by duration | 6 months after alloHCT
Overall corticosteroid requirement for treatment of chronic GvHD as measured by dose | 6 months after alloHCT
Overall corticosteroid requirement for treatment of chronic GvHD as measured by duration | 12 months after alloHCT
Overall corticosteroid requirement for treatment of chronic GvHD as measured by dose | 12 months after alloHCT
Overall corticosteroid requirement for treatment of chronic GvHD as measured by dose | 24 months after alloHCT
Overall corticosteroid requirement for treatment of chronic GvHD as measured by duration | 24 months after alloHCT
Necessity to use alternative treatment modalities for chronic GvHD | 6 months after alloHCT
  -The use of additional systemic immune suppressive agents will be captured at each study visit.
Necessity to use alternative treatment modalities for chronic GvHD | 12 months after alloHCT
  -The use of additional systemic immune suppressive agents will be captured at each study visit.
Necessity to use alternative treatment modalities for chronic GvHD | 24 months after alloHCT
  -The use of additional systemic immune suppressive agents will be captured at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Iskra Pusic, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu